CLINICAL TRIAL: NCT02547779
Title: Isotonic Solutions and Major Adverse Renal Events Trial in Non-Medical Intensive Care Units
Brief Title: Isotonic Solutions and Major Adverse Renal Events Trial in the Non-Medical Intensive Care Unit (SMART-SURG)
Acronym: SMART-SURG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Todd Rice, Associate Professor of Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB# 141349
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Results first posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Critical Illness; Acute Kidney Injury
Keywords: crystalloid; acute kidney injury
MeSH Terms: conditions — Critical Illness; Acute Kidney Injury | interventions — Saline Solution; Sodium Chloride; Ringer's Lactate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.9% Saline (Active Comparator): Patients in an ICU block randomized to physiologically-balanced isotonic fluid will receive 0.9% Saline whenever isotonic intravenous fluid administration is ordered by the treating provider.
  Interventions: Other: 0.9% Saline
- Physiologically-balanced (Active Comparator): Patients in an ICU block randomized to physiologically-balanced isotonic fluid will receive Plasma-Lyte© A or Lactated Ringer's whenever isotonic intravenous fluid administration is ordered by the treating provider.
  Interventions: Other: Physiologically-balanced isotonic crystalloid

INTERVENTIONS:
Other: 0.9% Saline — 0.9% Saline will be used whenever an isotonic crystalloid is ordered
  Other Names: Normal Saline; 0.9% sodium chloride
  Arms: 0.9% Saline
Other: Physiologically-balanced isotonic crystalloid — Lactated Ringers or Plasma-Lyte© A will be used whenever an isotonic crystalloid is ordered
  Other Names: Lactated Ringers; Ringer's Lactate; Plasma-Lyte© A
  Arms: Physiologically-balanced

SUMMARY:
The administration of intravenous fluids is ubiquitous in the care of the critically ill. Commonly available isotonic crystalloid solutions contain a broad spectrum electrolyte compositions including a range chloride concentrations. Recent studies have associated solutions with supraphysiologic chloride content with hyperchloremia, metabolic acidosis and renal vasoconstriction, acute kidney injury and renal replacement therapy, and increased mortality but no large, randomized-controlled trials have been conducted. SMART-SURG will be a large, cluster-randomized, multiple-crossover trial enrolling critically ill patients from the non-medical ICUs at Vanderbilt University from October 2015 until April 2017. The primary endpoint will be the incidence of Major Adverse Kidney Events in 30 days after enrollment (MAKE30 is the composite of death, new renal replacement, or persistent renal dysfunction at discharge).

DETAILED DESCRIPTION:
SMART-SURG is a large, cluster-randomized, multiple-crossover trial of 0.9% saline versus physiologically-balanced isotonic crystalloids (Lactated Ringers or Plasma-Lyte© A) with regard to the incidence of major adverse kidney events by 30 days in patients admitted to non-medical intensive care units. All patients admitted to participating non-medical intensive care units at Vanderbilt University medical center who are 18 years or older will be enrolled. The study will occur in one-month blocks. Each participating ICU will be randomized to an initial fluid group (0.9% saline or physiologically balanced isotonic crystalloids). The assigned fluid will be used exclusively for all patients receiving isotonic crystalloid for the duration of the month-long block (except in the presence of pre-specified contraindications). The assigned study fluid will switch at the end of each month-long block such that half of the months are assigned to 0.9% saline and half of the months to physiologically balance fluid. The primary endpoint will be major adverse kidney events by 30 days (MAKE30 is the composite of death, new renal replacement therapy, or persistent renal dysfunction at discharge). All aspects of study design, intervention, and data collection will be harmonized with an ongoing, independent study addressing the same question in the medical intensive care unit at Vanderbilt University during a similar study period (SMART-MED). A pre-specified data analysis plan will dictate the harmonized analysis of SMART-MED and SMART-SURG.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to a participating non-medical intensive care unit (ICU) at Vanderbilt University Medical Center

Exclusion Criteria:

* Age<18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10421 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd W Rice, MD, MSc, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Finfer S, Liu B, Taylor C, Bellomo R, Billot L, Cook D, Du B, McArthur C, Myburgh J; SAFE TRIPS Investigators. Resuscitation fluid use in critically ill adults: an international cross-sectional study in 391 intensive care units. Crit Care. 2010;14(5):R185. doi: 10.1186/cc9293. Epub 2010 Oct 15. PMID 20950434
- [Background] Yunos NM, Kim IB, Bellomo R, Bailey M, Ho L, Story D, Gutteridge GA, Hart GK. The biochemical effects of restricting chloride-rich fluids in intensive care. Crit Care Med. 2011 Nov;39(11):2419-24. doi: 10.1097/CCM.0b013e31822571e5. PMID 21705897
- [Background] Yunos NM, Bellomo R, Hegarty C, Story D, Ho L, Bailey M. Association between a chloride-liberal vs chloride-restrictive intravenous fluid administration strategy and kidney injury in critically ill adults. JAMA. 2012 Oct 17;308(15):1566-72. doi: 10.1001/jama.2012.13356. PMID 23073953
- [Derived] Lombardo S, Smith MC, Semler MW, Wang L, Dear ML, Lindsell CJ, Freundlich RE, Guillamondegui OD, Self WH, Rice TW; Isotonic Solutions and Major Adverse Renal Events Trial (SMART) Investigators and Vanderbilt Learning Healthcare System Platform Investigators. Balanced Crystalloid versus Saline in Adults with Traumatic Brain Injury: Secondary Analysis of a Clinical Trial. J Neurotrauma. 2022 Sep;39(17-18):1159-1167. doi: 10.1089/neu.2021.0465. PMID 35443809
- [Derived] Semler MW, Self WH, Wanderer JP, Ehrenfeld JM, Wang L, Byrne DW, Stollings JL, Kumar AB, Hughes CG, Hernandez A, Guillamondegui OD, May AK, Weavind L, Casey JD, Siew ED, Shaw AD, Bernard GR, Rice TW; SMART Investigators and the Pragmatic Critical Care Research Group. Balanced Crystalloids versus Saline in Critically Ill Adults. N Engl J Med. 2018 Mar 1;378(9):829-839. doi: 10.1056/NEJMoa1711584. Epub 2018 Feb 27. PMID 29485925
- [Derived] Semler MW, Self WH, Wang L, Byrne DW, Wanderer JP, Ehrenfeld JM, Stollings JL, Kumar AB, Hernandez A, Guillamondegui OD, May AK, Siew ED, Shaw AD, Bernard GR, Rice TW; Isotonic Solutions and Major Adverse Renal Events Trial (SMART) Investigators; Pragmatic Critical Care Research Group. Balanced crystalloids versus saline in the intensive care unit: study protocol for a cluster-randomized, multiple-crossover trial. Trials. 2017 Mar 16;18(1):129. doi: 10.1186/s13063-017-1871-1. PMID 28302179

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Isotonic Solutions and Major Adverse Events Trial (SMART) was registered for the medical ICU (NCT02444988), which enrolled 5381 patient beginning on June 1 2015, and then for the surgical ICUs (NCT02547779), which enrolled 10,421 patients beginning on October 1 2015. The overall SMART trial enrolled 15,802 patients and ended on April 30 2017.
Groups:
- 0.9% Sodium Chloride: Patients in an ICU block randomized to saline will receive 0.9% sodium chloride whenever isotonic intravenous crystalloid administration is ordered by the treating provider.
  Saline: 0.9% sodium chloride will be used whenever an isotonic crystalloid is ordered
- Balanced Crystalloids: Patients in an ICU block randomized to balanced crystalloids will receive Plasma-Lyte A or Lactated Ringer's whenever isotonic intravenous crystalloid administration is ordered by the treating provider.
  Balanced crystalloid: Lactated Ringers or Plasma-Lyte A will be used whenever an isotonic crystalloid is ordered
Period: Overall Study
Arm/Group | 0.9% Sodium Chloride | Balanced Crystalloids
Started | 5214 | 5207
Completed | 5214 | 5207
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.9% Sodium Chloride | Balanced Crystalloids | Total
Number analyzed (Participants) | 5214 | 5207 | 10421
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [44 to 69] | 57 [44 to 69] | 57 [44 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2052 | 2108 | 4160
  Male | 3162 | 3099 | 6261
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4344 | 4352 | 8696
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 870 | 855 | 1725

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Kidney Event Within 30 Days
Description: The primary outcome was the proportion of patients who met one or more criteria for a major adverse kidney event within 30 days - the composite of death, new receipt of renal-replacement therapy, or persistent renal dysfunction (defined as a final inpatient creatinine value ≥200% of the baseline value) - all censored at hospital discharge or 30 days after enrollment, whichever came first.
Time Frame: 30 days after enrollment censored at hospital discharge
Population: Of 15,802 patients in the SMART trial, 7,860 were assigned to saline and 7,942 were assigned to balanced crystalloids, of whom 10,421 were enrolled to surgical ICUs with 5,214 assigned to saline and 5,207 assigned to balanced crystalloids.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.9% Sodium Chloride | Balanced Crystalloids
Number analyzed (Participants) | 5214 | 5207
Participants | 551 | 524
Statistical Analysis 1: Comparison: 0.9% Sodium Chloride vs Balanced Crystalloids; Test type: Superiority; p < 0.05, Regression, Logistic; Odds Ratio (OR) = 0.95

2. Secondary Outcome: 30-day In-hospital Mortality
Description: Death before hospital discharge, censored at 30 days after enrollment
Time Frame: 30 days after enrollment censored at hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | 0.9% Sodium Chloride | Balanced Crystalloids
Number analyzed (Participants) | 5214 | 5207
Participants | 408 | 400
Statistical Analysis 1: Comparison: 0.9% Sodium Chloride vs Balanced Crystalloids; Test type: Superiority; p < 0.05, Regression, Logistic; Odds Ratio (OR) = 0.98

ADVERSE EVENTS:
Time Frame: 30 days
Description: An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation participant administered an intervention that does not necessarily have to have a causal relationship with this treatment. An adverse event therefore can be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an intervention, whether or not the incident is considered to be related to the intervention.
Arm/Group | 0.9% Sodium Chloride | Balanced Crystalloids
All-Cause Mortality (participants affected / at risk) | 408/5214 | 400/5207
Serious Adverse Events (participants affected / at risk) | 0/5214 | 0/5207
Other Adverse Events (participants affected / at risk) | 0/5214 | 1/5207
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.9% Sodium Chloride (N=5214) | Balanced Crystalloids (N=5207)
Adverse Event (Renal and urinary disorders) | 0 (0) | 1 (1) — Patient received Plasma-Lyte A® as post-filter replacement fluid during continuous RRT instead of 0.9% sodium chloride. The patient experience no significant changes in heart rate, systolic blood pressure, vasopressors, electrolytes or acid-base.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/79/NCT02547779/Prot_SAP_000.pdf